CLINICAL TRIAL: NCT05531227
Title: Corticosteroid Therapy for Persistent Synovitis in Acute Septic Arthritis on Native Joint
Acronym: SYNOVITIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8654
Record Dates: First submitted 2022-06-08; First posted 2022-09-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-06

CONDITIONS: Arthritis, Septic
Keywords: Arthritis, Septic; synovitis; Corticosteroid therapy; Inflammatory response; Native joint
MeSH Terms: conditions — Arthritis, Infectious; Synovitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute septic arthritis is a rare but life-threatening and functionally serious disease. The improvement or disappearance of pain and functional recovery are sometimes difficult to obtain, with in some cases the persistence of synovitis due to a prolonged local inflammatory response, despite early and effective treatment. The consequences are significant for patients with often significant chronic pain, repercussions on autonomy and/or profession. An unfavorable evolution with joint destruction and need for replacement by a prosthesis is not uncommon.

Corticosteroid therapy is widely used in rheumatology in similar tables, for the purpose of drug synovectomy, with good results. The risk of infection remains the main contraindication to its use.

There are very few studies on its use in septic arthritis, either fundamentally or in humans, for which there are no data in adults. However, these have shown results encouraging the investigators not to neglect this therapy.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* having presented with septic arthritis and treated at the Strasbourg University Hospital between January 1, 2012 and December 31, 2021
* clinical finding of persistent synovitis, defined by the presence of pain, effusion or joint stiffness despite well-conducted treatment
* having had a diagnosis of joint infection proven by a positive culture of the joint fluid to a pathogenic germ
* having had treatment with local or systemic corticosteroids.

Exclusion criteria:

* Patient who has expressed his opposition to the reuse of his data for scientific research purposes.
* Absence of corticosteroid treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) having presented with septic arthritis and treated at the Strasbourg University Hospital between January 1, 2012 and December 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12-13 (Estimated); Study Completion 2023-12-13 (Estimated)

PRIMARY OUTCOMES:
Complete regression of the pain in a fast way | 6 months after treatment with corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Jeannot GAUDIAS, MD, Principal Investigator — Service de Chirurgie Orthopédique Septique - CHU de Strasbourg - France
Locations (1):
- Service de Chirurgie Orthopédique Septique - CHU de Strasbourg - France, Strasbourg, France